CLINICAL TRIAL: NCT03921983
Title: Non Invasive Evaluation of Muscle Hypoxia in Chronic Obstructive Pulmonary Disease Patient
Brief Title: Non Invasive Evaluation of Muscle Hypoxia in COPD Patient (EVANIMUS)
Acronym: EVANIMUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RBHP 2018 COSTES; 2018-A02206-49 (Other: 2018-A02206-49)
Record Dates: First submitted 2019-04-15; First posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease); Hypoxemia
Keywords: muscle oxygenation; hypoxia; mitochondrial function; non invasive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypoxia

STUDY DESIGN:
Intervention Model Description: measurements will be made with and without short term oxygen supplementation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LTOT + (Experimental): COPD patients with long term oxygenotherapy
  Interventions: Other: Oxygen supplementation
- LTOT - (Active Comparator): COPD patients without chronic hypoxemia (no LTOT)
  Interventions: Other: Oxygen supplementation

INTERVENTIONS:
Other: Oxygen supplementation — short term O2 supplementation during 1 hour

SUMMARY:
Peripheral muscle oxidative function is altered in COPD(chronic obstrutive pulmonary disease) patients. Multiple factors could contribute to this dysfunction including chronic hypoxia and deconditioning (sedentarity).

The evaluation of mitochondrial function is based on invasive method (muscle biopsy and in vitro respirometry) or magnetic resonance spectroscopy limited to small muscle groups. Recently, a non invasive method has been described using Near InfraRed Spectroscopy (NIRS). During arterial occlusion, muscle deoxygenation is only dependent of local oxygen consumption. The time constant recovery (k) of the deoxygenation during repeated ischemia periods has been shown to be correlated to measurements of maximal mitochondrial capacity.

k is lower in COPD patients compared to smokers without bronchial obstruction. However, the influence of arterial hypoxia has never been studied precisely, no more than the confounding effect of deconditioning on k.

So , the aim is to compare k in COPD patients with chronic hypoxemia (treated with long term oxygenotherapy, LTOT+ group) and patients without hypoxia, matched for their physical activity (LTOT- group).

The hypothe is that k will be lower in LTOT+ group compared to LTOT- group and that short term O2 supplementation will improve it, which would suggest a muscle hypoxia. By contrast, O2 should not influence k in LOT- group, in whom it is mainly determined by muscle conditioning.

DETAILED DESCRIPTION:
Investigator will compare mVO2 time constant in 2 groups of COPD (chronic obstrutive pulmonary disease) patients matched for age, sex, physical activity (estimated by GPAQ questionnaire (Global Physical Activity Questionnaire)), one with chronic hypoxemia (LTOT+ group) and one without blood gas abnormalities (LTOT- group)..

Inclusion visit It will allow to calculate physical activity in Mets.min/week, from the GPAQ questionnaire. The patient will also be accustomed to the repeated arterial occlusion procedure. A pneumatic cuff will be wrapped around the thigh and will be progressively inflated to a suprasystolic value (rapid air inflation system Hokanson), from 160 mmHg up to tolerated maximal pressure (max 220 mmHg).

Experimental visit

* Muscle biopsy. A biopsy of the vastus lateralis will be performed while breathing ambient air. After disinfection and anesthesia of skin and subcutaneous tissue, an automatic biopsy gun (Monopty Bard 14G) will be introduced in the muscle and a 20 mg biopsy will be withdrawn. The maximal mitochondrial O2 consumption and mitochondrial affinity for O2 will be immediately measured with high resolution respirometry (Oroboros, 10 mg tissue). A 10 mg fragment will be stored in liquid nitrogen for mRNA analysis of hypoxia driven genes (Hypoxia-inducible Factor 1, Vascular Endothelial Growth Factor, Carbonic Anhydrase 9, Heme Oxygenase 1).
* mVO2 time constant measurement (k, min-1) in ambient air. A NIRS probe (Oxymon III) will be placed on the thigh (contralateral to the muscle biopsy) and secured with an elastic wrap. The NIRS signal will be displayed continuously and recorded on a software (Oxysoft) The inflation cuff will be placed upstream the NIRS probe. After 5 to 10 isometric contractions of the quadriceps, the cuff will be rapidly inflated (maximal tolerated pressure determined during the inclusion visit) and deflated according to a predetermined protocol: 5 s /5 s 5 times, followed by 7 s /7 s 5 times and then 10 s/10 s 10 times. The deoxygenation kinetics (% deoxygenation/min) will be calculated for every occlusion and these deoxygenation indices will be expressed over time in order to calculate the time constant of the exponential relationship (k, min-1). This sequence will be repeated twice and the k values will be averaged.
* mVO2 time constant measurement with O2. Oxygen therapy will be given to the patient for 1 hour before repeating the k determination as described above. Oxygen flow will be set to the habitual flow rate in the LTOT+ group, and an arbitrary 3 L/min flow rate in the LTOT- group.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnostic
* Both sex
* 18 <Age <80 years old
* LTOT- group : PaO2 ≥ 65 mmHg and SaO2≥ 92%
* LTOT+ group: long term oxygenotherapy prescribed for more than 3 months, with daily use between 12 and 15 hours.

Patients in both groups will be matched for age (± 5 years), sex and physical activity estimated by GPAQ questionnaire (± 15% Mets.min/week).

Exclusion Criteria:

* Recent cardiorespiratory exacerbation (<6 weeks).
* Pulmonary rehabilitation program during the last 2 months
* Continuous LTOT (24 hours) or deambulation O2 therapy alone
* Anticoagulant drugs
* Hematocrit outside the normal range (35-50%)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
mVO2 recovery time constant (k) measured while breathing ambient air | day 1
  Time constant (min-1) of NIRS muscle oxygenation kinetics following repetitive arterial occlusions

SECONDARY OUTCOMES:
variation of k with oxygen supplementation | day 1
  Difference of the time constant (k, min-1) between 2 conditions: ambient air and with oxygen supplementation
Mitochondrial affinity for O2 | day 1
  Apparent K (µmol O2/min/g tissue) measured with respirometry on permeabilized muscle fibers at decreasing concentration of O2

CONTACTS AND LOCATIONS:
Overall Officials: Frédériv Costes, MD, PhD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France